CLINICAL TRIAL: NCT04738422
Title: Determining Airway pH by Compartmental Exhaled Nitric Oxide Levels During Alkaline Buffer Challenge
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael D. Davis, Assistant Research Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003838272
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Airway Disease
MeSH Terms: interventions — Optate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alkaline glycine Inhalation (Experimental): Subjects inhale alkaline glycine
  Interventions: Drug: Alkaline glycine

INTERVENTIONS:
Drug: Alkaline glycine — Subjects will inhale alkaline glycine via nebulizer. Alkaline glycine is an alkaline medication designed for medication.
  Other Names: Optate

SUMMARY:
Airway pH imbalances cause numerous adverse physiological changes within the airways, including hyperreactivity, cough, bronchoconstriction, ciliopathy, decreased response to bronchodilators, bacterial growth, nitrosative/oxidative stress, neutrophilic/eosinophilic inflammation, and cell death. Airway pH is known to be low (acidic) in chronic and acute pulmonary diseases. The gold standard approach to measuring airway pH is to bronchscopically obtain epithelial cell lining fluid using protected brush sampling. The expense and invasive nature of this approach is a barrier to fully characterizing the role of airway pH in the health and disease. In this study, we will evaluate non-invasive clinical methods that can be done using equipment standard in clinical pulmonary function laboratories for measuring airway pH.

DETAILED DESCRIPTION:
Airway pH imbalances cause numerous adverse physiological changes within the airways, including hyperreactivity, cough, bronchoconstriction, ciliopathy, decreased response to bronchodilators, bacterial growth, nitrosative/oxidative stress, neutrophilic/eosinophilic inflammation, and cell death. Airway pH is known to be low (acidic) in chronic and acute pulmonary diseases. The gold standard approach to measuring airway pH is to bronchscopically obtain epithelial cell lining fluid using protected brush sampling. The expense and invasive nature of this approach is a barrier to fully characterizing the role of airway pH in the health and disease. In this study, the investigator will evaluate non-invasive clinical methods that can be done using equipment standard in clinical pulmonary function laboratories for measuring airway pH.

The study team has previously demonstrated that exhaled breath condensate (EBC) pH and changes in fractional exhaled nitric oxide collected at 50mL/sec (FeNO50) after inhalation of an alkaline glycine buffer (AGB) indicate low airway pH. While EBC pH is the most common method and validated method for estimating airway pH, the investigators believes that the change in FeNO50 is the most sensitive test for general airway pH. Specifically, this proposed test makes use of the facts that the pH of nitrite/nitrous acid (NO2-/HNO2) is just under 4. Nitrous acid thus evolves nitric oxide (NO) when pH is less than 6.5, and NO evolution stops when pH is above 7. Because endogenous human airway NO2- levels are normally low μM, (32) NO2 protonation can be used as a noninvasive test for airway pH. Using the Henderson-Hasselbalch equation, the investigator can use these changes in NO to calculate pH. The investigator has now done studies with both inhaled phosphate buffer and AGB, both of which show that specific patients with asthma have a significant fall in FeNO50 following buffer inhalation. While FeNO50 is validated to represent the nitric oxide levels of the middle airways, sampling can be done at several different flowrates and times to evaluate the nitric oxide levels in different compartments of the lung. This can allow for regional airway pH measurement which would be helpful since many airway diseases are heterogeneous and regional. The investigator will further characterize the normal range of airway pH in health and disease compartmentally within the airways and in subsequent studies will evaluate the effects of clinically altering pH when it is abnormal.

It has been recently discovered that airway pH is integral to airway cell entry and replication of SARS-CoV-2 virus. Specifically, one of the pathways by which the virus enters cells and replicates is blocked by intracellular alkalinization. The investigator therefore tested to determine whether AGB would cause intracellular alkalinization in cultured primary human airway epithelial cells. It did; and the drug was well-tolerated by the cells in vitro (as it is in vivo).

The investigators believes that the next step is to determine whether AGB inhibits viral replication and viral entry in our primary human airway epithelial cultures. To do this, the investigator is partnering with the Indiana University BSL3 virology lab. The investigator has acquired the virus, completed preparations of it, and has infected human airway epithelial cultures with it. The study team is awaiting preliminary results of the effects of AGB on viral entry and replication. If in fact AGB inhibits viral cell entry and, thereby, replication, the investigator intends to expand the IND with the FDA, allowing a trial in patients at risk for respiratory distress associated with known COVID-2 respiratory disease. Ultimately, outcomes of this trial would be proposed to include: mortality (primary); as well as ICU length of stay and oxygen saturation index area under the curve (secondary). The investigator has submitted grants to the NIH, the DoD, and several other agencies for this project.

The study proposed here will not only provide further insight into the use of AGB in a larger population but also will allow for evaluation of airway pH in those receiving it which could be used to guide therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Study sample will consist of individuals aged 18-60 with a diagnosis of acute or chronic respiratory disorders or normal subjects with no pulmonary disease.

Healthy subjects may include:

1. Adult males or females age ≥ 18 and ≤ 60 years at time of enrollment
2. Non-smokers
3. Person with no history of asthma, chronic obstructive pulmonary disease (COPD), or other chronic lung disease
4. Person with no history of severe allergic/atopic disease requiring immunotherapy or immunomodulators

Subjects with pulmonary disease may include:

1. Person with well-documented disease with objective diagnostics such a lung function or genetic testing.
2. Person with FEV1 > 55% predicted on the day of study procedures.
3. Person who is clinically stable with no significant changes in health status within 4 weeks.

Exclusion Criteria:

* • Subjects that are mechanically ventilated.

  * Subjects that are unable or unwilling to cooperate with specimen collection.
  * Subjects with diagnosis of any medical condition that in the investigator's opinion would make them unsuitable for study participation.
  * Subjects who experienced a pulmonary exacerbation within the 4 weeks prior to visit.
  * Subjects requiring continuous oxygen therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Compartmental FeNO | Study is a single visit, lasting less than two hours
  Measuring compartmental FeNO before inhaled alkaline glycine and after inhaled alkaline glycine
Calculated compartmental airway pH | Study is a single visit, lasting less than two hours
  Calculating compartmental FeNO before inhaled alkaline glycine and after inhaled alkaline glycine
Exhaled Breath Condensate (EBC) pH | Study is a single visit, lasting less than two hours
  Measuring the pH of EBC before and after inhaled alkaline glycine

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States